CLINICAL TRIAL: NCT00815698
Title: Effect of Suture for Mesh Fixation in Lichtenstein Hernia Repair, a Prospective Controlled Randomized Trial
Brief Title: Effect of Suture for Mesh Fixation in Lichtenstein Hernia Repair
Acronym: Dangrip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob Rosenberg (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Frederikshavn Hospital (Unknown); Nyborg Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Jacob Rosenberg, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPODenmark001
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Inguinal Hernia
Keywords: pain
MeSH Terms: conditions — Hernia, Inguinal; Pain | interventions — Sutures; Polypropylenes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- no suture (Active Comparator): self-adhesive mesh, i.e. no suture for mesh fixation
  Interventions: Procedure: no suture
- Suture (Experimental): Suture for mesh fixation
  Interventions: Procedure: suture

INTERVENTIONS:
Procedure: suture — suture for mesh fixation
  Other Names: Prolene and Vicryl sutures
  Arms: Suture
Procedure: no suture — no suture for mesh fixation, because we use a self-adhesive mesh
  Other Names: Progrip mesh
  Arms: no suture

SUMMARY:
The investigators want to evaluate the effect of suturing the mesh versus using a self-adhesive mesh for Lichtenstein hernia repair. Effect parameters include chronic pain.

DETAILED DESCRIPTION:
Pain is a frequent problem after open inguinal hernia repair. The most frequent operative technique for inguinal hernia repair in adults is the Lichtenstein mesh repair, where a polypropylene mesh is sutured to the tissue in the inguinal region. We therefore want to evaluate the effect of suture for mesh fixation on the occurrence of chronic pain 12 months after operation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males 18-80 years
* Primary inguinal unilateral hernia

Exclusion Criteria:

* Recurrent hernia
* Bilateral, scrotal or femoral hernia
* BMI above 35

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, MD, DSc, Principal Investigator — Herlev Hospital
Locations (5):
- Denmark (5):
  - Bispebjerg Hospital, Copenhagen, Copenhaven
  - Frederikshavn Hospital, Frederikshavn, Frederikshavn
  - Gentofte Hospital, Gentofte Municipality, Hellerup
  - Randers Hospital, Randers, Randers
  - Nyborg Hospital, Nyborg, Svendborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jorgensen LN, Sommer T, Assaadzadeh S, Strand L, Dorfelt A, Hensler M, Rosenberg J; Danish Multicentre DANGRIP Study Group. Randomized clinical trial of self-gripping mesh versus sutured mesh for Lichtenstein hernia repair. Br J Surg. 2013 Mar;100(4):474-81. doi: 10.1002/bjs.9006. Epub 2012 Nov 30. PMID 23203909
- [Derived] Rosenberg J, Henriksen NA, Jorgensen LN. Multicenter data acquisition made easy. Trials. 2010 Apr 30;11:49. doi: 10.1186/1745-6215-11-49. PMID 20433715

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | no Suture | Suture
Started | 163 | 171
Completed | 163 | 171
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Suture | Suture | Total
Number analyzed (Participants) | 163 | 171 | 334
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.8 [40.2 to 65.1] | 59.9 [45.8 to 67.5] | 58.0 [40.2 to 67.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 163 | 171 | 334
Region of Enrollment [Number; unit: participants]
  Denmark | 163 | 171 | 334

OUTCOME MEASURES:

1. Primary Outcome: Pain, Numbness and Discomfort in the Groin
Description: The primary endpoint was a combined measure that evaluated the prevalence of symptoms considered moderate or severe. These symptoms included moderate to severe chronic pain and/or numbness and/or groin discomfort at the 12-month visit.
Time Frame: 12 months after surgery
Measure: Number; unit: participants
Arm/Group | no Suture | Suture
Number analyzed (Participants) | 163 | 171
participants | 28 | 34

2. Secondary Outcome: Recurrence
Description: recurrence means recurrence of the hernia defined as a new lump in the inguinal region diagnosed by a surgeon to be a new inguinal hernia.
Time Frame: 12 months after surgery
Measure: Number; unit: participants
Arm/Group | no Suture | Suture
Number analyzed (Participants) | 163 | 171
participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | no Suture | Suture
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/171
Other Adverse Events (participants affected / at risk) | 0/163 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes